CLINICAL TRIAL: NCT03562156
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oteseconazole (VT-1161) Oral Capsules in the Treatment of Subjects With Recurrent Vulvovaginal Candidiasis
Brief Title: A Study of Oral Oteseconazole for the Treatment of Patients With Recurrent Vaginal Candidiasis (Yeast Infection)
Acronym: VIOLET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mycovia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VMT-VT-1161-CL-011
Record Dates: First submitted 2018-06-01; First posted 2018-06-19 (Actual); Results first posted 2022-01-13 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Recurrent Vulvovaginal Candidiasis
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — VT-1161

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oteseconazole (VT-1161) 150mg capsule (Experimental): Once daily for 7 days starting at Day 1, followed by once weekly for 11 weeks
  Interventions: Drug: Oteseconazole (VT-1161)
- Placebo capsule (Placebo Comparator): Once daily for 7 days starting at Day 1, followed by once weekly for 11 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oteseconazole (VT-1161) — Oteseconazole (VT-1161) 150mg capsule
  Arms: Oteseconazole (VT-1161) 150mg capsule
Drug: Placebo — matching placebo capsule
  Arms: Placebo capsule

SUMMARY:
Recurrent vulvovaginal candidiasis (RVVC), also known as recurrent yeast infections, is defined as at least 3 episodes of acute VVC in the past 12 months. Several properties of oteseconazole (VT-1161) suggest that it might be a safer and more effective treatment for RVVC than other oral anti-fungal medicines.

This study will evaluate the effectiveness and safety of oteseconazole (VT-1161) for the treatment of RVVC and consists of 2 parts. The first part of the study is a 2-week period for the treatment of the patient's current VVC episode with 3 150mg doses of fluconazole. The 2nd part consists of 12 weeks, when the patient will take either oteseconazole (VT-1161) 150 mg or a placebo (according to a random assignment), and then a 36-week follow-up period.

In addition, at participating sites, an amendment to the study allows US patients who complete the initial 48 weeks without experiencing a confirmed RVVC episode to continue in a 48-week observational extension period designed to evaluate the continued effectiveness of oteseconazole (VT-1161).

This study is identical to VMT-VT-1161-CL-012 (NCT03561701).

ELIGIBILITY:
Key Inclusion Criteria:

* 3 or more episodes of acute VVC in the past 12 months
* Positive KOH or Gram stain
* Total vulvovaginal signs and symptoms score of ≥3 at screening visit
* Total vulvovaginal signs and symptoms score of <3 at baseline visit
* Must be able to swallow pills

Key Exclusion Criteria:

* Presence or a history of another vaginal or vulvar condition(s)
* Evidence of major organ system disease
* History of cervical cancer
* Poorly controlled diabetes mellitus
* Pregnant
* Recent use of topical or systemic antifungal or antibacterial drugs
* Recent use of immunosuppressive or systemic corticosteroid therapies

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2021-08-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - 31123, Birmingham, Alabama
  - 31108, San Diego, California
  - 31139, Lauderdale Lakes, Florida
  - 31143, Sarasota, Florida
  - 31106, Wellington, Florida
  - 31111, Norcross, Georgia
  - 31146, Covington, Louisiana
  - 31107, Metairie, Louisiana
  - 31105, Metairie, Louisiana
  - 31147, Fall River, Massachusetts
  - 31118, Las Vegas, Nevada
  - 31103, Las Vegas, Nevada
  - 31114, Lawrenceville, New Jersey
  - 31142, Port Jefferson, New York
  - 31127, West Seneca, New York
  - 31132, Greensboro, North Carolina
  - 31116, Morehead City, North Carolina
  - 31144, Raleigh, North Carolina
  - 31145, Winston-Salem, North Carolina
  - 31125, Franklin, Ohio
  - 31134, Philadelphia, Pennsylvania
  - 31120, Bristol, Tennessee
  - 31102, Houston, Texas
  - 31117, Draper, Utah
  - 31113, Richmond, Virginia

REFERENCES:
- [Derived] Sobel JD, Donders G, Degenhardt T, Person K, Curelop S, Ghannoum M, Brand SR. Efficacy and Safety of Oteseconazole in Recurrent Vulvovaginal Candidiasis. NEJM Evid. 2022 Aug;1(8):EVIDoa2100055. doi: 10.1056/EVIDoa2100055. Epub 2022 Jul 26. PMID 38319878
- [Derived] Vanreppelen G, Nysten J, Baldewijns S, Sillen M, Donders G, Van Dijck P. Oteseconazole (VIVOJA) for prevention of recurrent vulvovaginal candidiasis. Trends Pharmacol Sci. 2023 Jan;44(1):64-65. doi: 10.1016/j.tips.2022.10.004. Epub 2022 Nov 14. No abstract available. PMID 36396498

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 438 subjects were enrolled in a 2-week Induction Phase after providing consent. During the Induction Phase, subjects received 3 sequential 150mg of fluconazole administered 72 hours apart. Subjects whose presenting acute VVC (vulvovaginal candidiasis) episode resolved during the Induction Phase (a total of 326) entered a 48-week Maintenance Phase comprised of a 12-week treatment period and a 36-week follow-up period.
Groups:
- Oteseconazole (VT-1161): 1 oteseconazole 150mg capsule once daily for 7 days starting at Day 1, then once weekly for 11 weeks
- Placebo: 1 placebo capsule once daily for 7 days starting at Day 1, then once weekly for 11 weeks
Period: Overall Study
Arm/Group | Oteseconazole (VT-1161) | Placebo
Started | 217 | 109
Completed | 182 | 91
Not Completed | 35 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oteseconazole (VT-1161) | Placebo | Total
Number analyzed (Participants) | 217 | 109 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10.3) | 34 (9.9) | 34 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 109 | 326
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 33 | 12 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 17 | 43
  White | 156 | 80 | 236
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 85 | 39 | 124
  Bulgaria | 50 | 23 | 73
  Canada | 8 | 8 | 16
  Japan | 32 | 12 | 44
  Poland | 33 | 24 | 57
  United Kingdom | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With 1 or More Culture-Verified Acute VVC Episodes During the Maintenance Phase of the Study in the Intent-to-Treat Population
Description: The primary efficacy outcome measure was the percentage of subjects with 1 or more culture-verified acute VVC episodes during the maintenance phase (post-randomization through Week 48) in the intent-to-treat population. An acute VVC episode during the maintenance phase (considered a recurrent episode) was defined as a positive fungal culture for Candida species and a clinical signs and symptoms score of ≥3. To calculate the signs and symptoms score, each vulvovaginal sign (erythema, edema, excoriation) and symptom (itching, burning, irritation) was scored using the following scale, with a higher score indicating a worse outcome.
  0 = none (complete absence of any sign or symptom), 1 = mild (slight), 2 = moderate (definitely present), 3 = severe (marked, intense)
Time Frame: Maintenance phase (post-randomization through Week 48)
Population: Analysis was performed on the ITT population which included all randomized subjects. Missing values were imputed with multiple imputation using the following auxiliary information: region, treatment, baseline body mass index, baseline age, ethnicity, and visit.
Measure: Number; unit: percentage of subjects
Arm/Group | Oteseconazole (VT-1161) | Placebo
Number analyzed (Participants) | 217 | 109
percentage of subjects | 6.7 | 42.8

ADVERSE EVENTS:
Time Frame: Day 1 through Week 48
Description: The safety population was defined as all randomized subjects who received at least 1 dose of investigational product, which was not administered until Day 1. Treatment-emergent adverse events were defined as adverse events that occurred after the subject received her initial dose of investigational product. Adverse event data were not collected during the induction phase.
Arm/Group | Oteseconazole (VT-1161) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/217 | 0/109
Serious Adverse Events (participants affected / at risk) | 3/217 | 3/109
Other Adverse Events (participants affected / at risk) | 129/217 | 63/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oteseconazole (VT-1161) (N=217) | Placebo (N=109)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal haemmorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oteseconazole (VT-1161) (N=217) | Placebo (N=109)
Nasopharyngitis (Infections and infestations) | 26 (37) | 7 (10)
Bacterial vaginosis (Infections and infestations) | 14 (19) | 11 (15)
Urinary tract infection (Infections and infestations) | 12 (14) | 7 (9)
Upper respiratory tract infection (Infections and infestations) | 9 (9) | 7 (7)
Sinusitis (Infections and infestations) | 12 (13) | 3 (3)
Cystitis (Infections and infestations) | 4 (6) | 8 (13)
Influenza (Infections and infestations) | 7 (7) | 1 (1)
Genital herpes (Infections and infestations) | 7 (8) | 0 (0)
Bronchitis (Infections and infestations) | 4 (6) | 2 (2)
Chlamydial infection (Infections and infestations) | 4 (5) | 2 (2)
Pharyngitis (Infections and infestations) | 6 (6) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 2 (3)
Vulvovaginal candidiasis (Infections and infestations) | 1 (2) | 2 (2)
Vulvitis (Infections and infestations) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 8 (10) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 3 (4)
Abdominal pain lower (Gastrointestinal disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 7 (7) | 2 (4)
Metrorrhagia (Reproductive system and breast disorders) | 5 (7) | 3 (3)
Menorrhagia (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 4 (5)
Headache (Nervous system disorders) | 8 (8) | 8 (10)
Acne (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (6)
Blood creatine phosphokinase increased (Investigations) | 7 (8) | 3 (3)
Pyrexia (General disorders) | 5 (5) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither institution nor investigator can disclose information pertaining to study until sponsor issues multi-center publication. If multi-center publication is not issued within 18 months of study completion and database lock at all sites, sponsor has 30 days from receipt to review institution's and/or investigator's communication and can require removal of confidential information other than study data and/or delay release of institution's and/or investigator's communication for 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT03562156/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-25): https://cdn.clinicaltrials.gov/large-docs/56/NCT03562156/SAP_001.pdf